CLINICAL TRIAL: NCT04622670
Title: Yoga Therapy During Chemotherapy and Radiation Treatment for Local-Regional Cervical Cancer
Brief Title: Yoga Therapy During Chemotherapy and Radiation Treatment for the Improvement of Physical and Emotional Well-Being in Patients With Stage IB2-IIIB Cervical Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0919; NCI-2020-02021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0919 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-04-30; First posted 2020-11-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB2 Cervical Cancer FIGO 2018; Stage IB3 Cervical Cancer FIGO 2018; Stage II Cervical Cancer FIGO 2018; Stage IIA Cervical Cancer FIGO 2018; Stage IIA1 Cervical Cancer FIGO 2018; Stage IIA2 Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (yoga group) (Experimental): Patients attend at least 2 yoga classes per week over 5-6 weeks lasting approximately 60 minutes each for up to 15 classes during the CRT. Patients also complete surveys pre-treatment, once a week, and post-treatment over and receive a yoga manual and DVD during and after CRT.
  Interventions: Other: Media Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Procedure: Yoga
- Group II (wait list control) (Active Comparator): Patients refrain from participating in any new stress management activities and receive a DVD. Patients are also offered 4 group yoga classes after 3 months of CRT. Patients also complete surveys as in Group I.
  Interventions: Other: Media Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Media Intervention — Receive DVD
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Procedure: Yoga — Attend yoga class
  Other Names: Yoga Therapy
  Arms: Group I (yoga group)

SUMMARY:
This trial studies how well yoga therapy works during chemotherapy and radiation treatment in improving physical and emotional well-being in patients with stage IB2-IIIB cervical cancer. Yoga therapy may help to balance the mind and body through exercise, meditation (focusing thoughts), and control of breathing and emotions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Establish feasibility of delivering a yoga therapy program during chemotherapy and radiation therapy (CRT) for loco-regionally advanced cervical cancer undergoing chemo-radiotherapy.

SECONDARY OBJECTIVES:

I. Measure the effects and variance of yoga on fatigue, depression, anxiety, pelvic pain and over-all quality of life (QOL) in cervical cancer (CxCa) patients undergoing primary treatment with CRT.

II. Examine changes in other psychosocial outcomes including ability to find meaning in the illness, spirituality and sexuality.

EXPLORATORY OBJECTIVE:

I. Evaluate whether markers of stress response (plasma levels of other pro-inflammatory cytokines, including interleukin-6 [IL-6], and IL-8, IL-10, VEGF, and CRP) change in response to yoga therapy and their association with fatigue, depression, anxiety, pelvic pain, meaning in the illness, experience, spirituality, and QOL in CxCa patients undergoing primary CRT.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (YOGA GROUP): Patients attend at least 2 yoga classes per week over 5-6 weeks lasting approximately 60 minutes each for up to 15 classes during the CRT. Patients also complete surveys pre-treatment, once a week, and post-treatment and receive a yoga manual and DVD during and after CRT.

GROUP II (WAIT LIST CONTROL): Patients refrain from participating in any new stress management activities and receive a DVD. Patients are also offered 4 group yoga classes after 3 months of CRT. Patients also complete surveys as in Group I.

ELIGIBILITY:
Inclusion Criteria:

* Score of =< 2 on Eastern Cooperative Oncology Group (ECOG) performance scale
* Able to speak English
* Federation of Gynecology and Obstetrics (FIGO) stage IB2 through IIIB biopsy-proven CxCa (adenocarcinoma, squamous cell carcinoma, and adenosquamous) with plan to undergo curative outpatient CRT at main campus MD Anderson Cancer Center

Exclusion Criteria:

* Medically documented restrictions at enrollment that could interfere with participation in the yoga interventions (i.e. uncontrolled vaginal bleeding)
* Medical illness that would prevent administration of full-dose chemotherapy
* Concurrent diagnosis of a second cancer
* Prior hysterectomy
* Neuroendocrine histology
* Patients who are pregnant

  * It is standard procedure to administer a pregnancy test before the start of CRT. Patients are deemed not pregnant by virtue of urine pregnancy test (UPT) or testing of the blood. Due to radiation and the nature of the disease, a patient becoming pregnant while on study is highly unlikely. In the event a patient were to get pregnant, they would be removed from study because their radiation therapy (RT) might be stopped or fetus would be terminated, which might influence other parameters that are being measured
* Patients with major psychiatric diagnoses (e.g., schizophrenia, bipolar disorder)
* Patients with extreme mobility issues, and
* Patients who have had a regular yoga practice (at least one time a month) in past 6 months prior to study enrollment or who are currently engaged in a regular mind-body practice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment to the yoga therapy protocol | Baseline up to 3 months post CRT
  90 patients will be screen to obtain at least 40 who are eligible and consent
Adherence to the yoga therapy protocol | Baseline up to 3 months post CRT
  At least 10 patients in the YG group must complete at least 50% of the required yoga sessions
Completion in the yoga therapy protocol | Baseline up to 3 months post CRT
  At least 25 of the 40 patients must complete any of the follow up measure between T3 and T5 in order to declare this study feasible

CONTACTS AND LOCATIONS:
Overall Officials: Lois M Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT04622670/ICF_000.pdf